CLINICAL TRIAL: NCT04287439
Title: Progressive Muscle Relaxation and Mindfulness Meditation on Neuropathic Pain, Fatigue and Quality of Life in Type 2 Diabetes Patients: A Randomized Clinical Trial
Brief Title: Relaxation and Meditation Techniques on Pain, Fatigue and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Nur Izgu, Assistant professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Neuropathy, Diabetic
Keywords: Fatigue, meditation, diabetic neuropathy, relaxation, quality of life.
MeSH Terms: conditions — Diabetic Neuropathies; Fatigue | interventions — Autogenic Training; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxation (Experimental): Patients will receive a training session for progressive muscle relaxation exercise.
  They will practice it daily at their home during 12 weeks. Patients will be called daily to ensure that patients perform the intervention according to the study protocol, and to assess their study-adherence.
  Interventions: Behavioral: Progressive muscle relaxation
- Meditation (Experimental): Patients will receive a training session for minfullness meditation They will practice it daily at their home during 12 weeks. Patients will be called daily to ensure that patients perform the intervention according to the study protocol, and to assess their study-adherence.
  Interventions: Behavioral: Mindfulness meditation
- Attention matched control group (Active Comparator): Patients will receive a training session focusing on the anatomy and physiological functions of the pancreas, general information about type 2 diabetes including signs, complication, and treatment methods.
  Interventions: Other: Attention matched control

INTERVENTIONS:
Behavioral: Progressive muscle relaxation — Patients will receive a training session for progressive muscle relaxation exercise They will practice it daily at their home during 12 weeks. Patients will be called daily to ensure that patients perform the intervention according to the study protocol, and to assess their study-adherence.
  Arms: Relaxation
Behavioral: Mindfulness meditation — Patients will receive a training session for mindfulness meditation. They will practice it daily at their home during 12 weeks. Patients will be called daily to ensure that patients perform the intervention according to the study protocol, and to assess their study-adherence.
  Arms: Meditation
Other: Attention matched control — Patients will receive a training session focusing on focusing on the anatomy and physiological functions of the pancreas, general information about type 2 diabetes including signs, complication, and treatment methods
  Arms: Attention matched control group

SUMMARY:
Patients with painful diabethic peripheral neuropathy will be entered.. Participants will be randomized to one of three study arms: Arm 1: relaxatio; Arm 2:meditation Arm 3: Attention matched control Hypothesis: Progressive muscle relaxation and mindfullness meditation will decrease severity of neuropathc pain and fatigue and improve quality of life.

DETAILED DESCRIPTION:
Previous reports have revealed that progressive muscle relaxation and meditation are promising for glycemic control in type 2 diabetes patients. On the other hand, research examining effects of these approaches on painful diabetic peripheral neuropathy, fatigue and quality of life is limited. The present study investigates the effects of progressive muscle relaxation and mindfullness meditation in a single-site, 3-arm, assessor blinded randomized, controlled study of 77 type 2 diabetes patients with painful diabetic peripheral neuropathy. Arm 1: relaxation; Arm 2: mindfulness meditation; Arm 3: Attention matched control. The investigators hypothesize that Progressive muscle relaxation and mindfulness meditation will decrease severity of neuropathic pain and fatigue and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with painful diabethic peripheral neuropathy ,
* being at least primary school graduates,
* not using any other complementary or integrative therapy during the study period

Exclusion Criteria:

* neuropathy history due to any other causes such as megaloblastic anemia, fibromyalgia, autoimmune diseases, hypothyroidism, and lumbar disc hernia
* having end-stage of renal failure, chronic obstructive pulmonary disease, advanced cardiac failure, musculoskeletal disorders or depression
* having a diabetic foot ulcer or amputation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
Change in pain severity | Baseline measurements, at the end of 12th week and two weeks after the completion of the interventions
  Pain severity will be measured based on patient report by a visual analog scale. Higher score means increase in pain severity.

SECONDARY OUTCOMES:
Change in fatigue severity | Baseline measurements, at the end of 12th week and two weeks after the completion of the interventions
  Fatigue severity will be measured based on patient report by the Functional Assessment of Chronic Illness- Fatigue Scale. Higher scores indicate that low level of fatigue.
Change in Quality of life status | baseline measurements, at the end of 12th week and two weeks after the completion of the interventions
  Quality of live will be measured by the Neuropathic Pain Impact on Quality of Life Questionnaire. Higher scores on the scale mean better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Izgu, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Ankara University Medical Faculty Ibni Sina Hospital Endocrinology Outpatient Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No